CLINICAL TRIAL: NCT04927832
Title: Detection of Small Fiber Neuropathies by the Non-invasive SUDOSCAN Method During Chronic Autoimmune Pathologies and / or Unexplained Pain Syndromes
Acronym: SUDOCU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-A01515-46
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Systemic Autoimmune Pathologies; Unexplained Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with chronic autoimmune pathology (Experimental)
  Interventions: Other: SUDOSCAN and EMG (electromyogram)
- Patients with unexplained pain syndrome (Experimental)
  Interventions: Other: SUDOSCAN and EMG (electromyogram)

INTERVENTIONS:
Other: SUDOSCAN and EMG (electromyogram) — The participants are evaluated clinically by a neurologist with evaluation by DN4 questionnaire, treatments and comorbidities (alcohol consumption, diabetes, etc.). They undergo from exploration by SUDOSCAN according to the already established methodology and an EMG

SUMMARY:
Very few studies have evaluated the prevalence of small fiber neuropathy (SFN) during pathologies that may be responsible for small fibers damage.

SUDOSCAN is a new rapid (2 minutes), automated, reproducible and non-invasive technology to assess small fiber neuropathy by sweat function.

With quantitative and reproducible results, SUDOSCAN allows physicians to early detect and follow-up peripheral neuropathy to monitor disease progression and assess treatment efficacy for a better patient management.

SUDOSCAN® could allow the identification of SFN in painful patients apart from another pathology already diagnosed responsible for SFN.

The purpose of the study SUDOCU is to assess the prevalence of small fiber neuropathies (SFN) in patients with systemic autoimmune pathologies or unexplained pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patient corresponding to one of the two following groups:

  1. Systemic autoimmune pathology known to be complicated by small fiber neuropathies.

     The following autoimmune pathologies will be included: Lupus, Sjogren, Scleroderma, Myositis, rheumatoid arthritis, Sarcoidosis, Vasculitis of small or medium vessels
  2. No conditions known to be responsible at SFN, unexplained pain symptoms
* Aged ≥ 18 years
* Having given free and informed written consent

Exclusion Criteria:

* Chronic alcoholism
* Unbalanced diabetes
* Chemotherapies
* HIV
* Vitamins B12, B1, B6 deficiencies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Percentage of patients presenting diagnosis of small fiber neuropathy in chronic pathologies and / or unexplained pain syndrome | 53 months

CONTACTS AND LOCATIONS:
Locations (1):
- BENNANI, Marseille, France

IPD SHARING:
Plan to Share IPD: No